CLINICAL TRIAL: NCT01511796
Title: Effectiveness of Botulinum Toxin Combined With Upper Limb Rehabilitation on Arm Function
Brief Title: Examining the Effectiveness of Combined Rehabilitation and Botulinum Toxin Injection on Functional Improvement of the Upper Limb After Stroke
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Parvin Eftekhar, principal inverstigator, Toronto Rehabilitation Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTul Rehab
Record Dates: First submitted 2012-01-06; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Stroke
Keywords: stroke; upper limb rehabilitation function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- upper limb rehabilitation for total of 6 months (Experimental): upper limb rehabiliation
  Interventions: Other: upper limb rehabiliation

INTERVENTIONS:
Other: upper limb rehabiliation — 3 months upper rehabilation (twice a week) and then 3 more months upper limb rehabitation ( twice a week)

SUMMARY:
The purpose of this study is to examine the effects of a combination of "Botulinum Toxin (BT) and Upper Limb (UL) rehabilitation" compared to "BT only" on UL motor function in adults with spasticity after stroke using a pre-post design. The research question is whether combination of BT and UL rehabilitation compared to BT only is more effective in improving the UL function, range of motion and pain.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* at least 4 months post stroke
* present with UL spasticity (MAS >1 in elbow and/or spasticity of the hand, wrist or shoulder)
* present with at lease a stage 3 of CMSA
* able to comply with the requirements of the protocol and UL therapy programme.

Exclusion Criteria:

* significant cognitive and speech impairments
* other upper limb impairments such as frozen shoulder
* another diagnosis which could contribute to upper limb spasticity .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth | up tp 2013

SECONDARY OUTCOMES:
Goal attaiment Scale | up tp 2013

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Rehabiliation institute, Toronto, Ontario, Canada